CLINICAL TRIAL: NCT07393269
Title: Accuracy of Implant Impression Techniques Using Scannable Healing Abutments Versus Conventional Methods. A Controlled Clinical Trial
Brief Title: Accuracy of Scannable Healing Abutments for Implant Impressions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sherif Aly Sadek (Other)
Responsible Party: Sponsor-Investigator, Sherif Aly Sadek, Associate Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 33-6-25
Record Dates: First submitted 2026-01-24; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Partially Edentulous Maxilla, Mandible
Keywords: Dental Impression Technique; Intraoral Scanning; Partial Edentulism; Digital Dentistry; Dental Implants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scannable Healing Abutment Digital Impression (Experimental): Intraoral digital impression using scannable healing abutments and an intraoral scanner.
  Interventions: Procedure: Digital implant impression using scannable healing abutments
- Open-Tray Conventional Impression (Active Comparator): Conventional splinted open-tray implant impression using polyvinyl siloxane.
  Interventions: Procedure: Open-tray implant impression
- Closed-Tray Conventional Impression (Active Comparator): Conventional closed-tray implant impression using polyvinyl siloxane.
  Interventions: Procedure: Closed-tray implant impression

INTERVENTIONS:
Procedure: Digital implant impression using scannable healing abutments — Digital acquisition of implant position using intraoral scanning of scannable healing abutments following second-stage surgery.
  Arms: Scannable Healing Abutment Digital Impression
Procedure: Open-tray implant impression — Conventional open-tray implant-level impression using splinted impression copings and polyvinyl siloxane material.
  Arms: Open-Tray Conventional Impression
Procedure: Closed-tray implant impression — Conventional closed-tray implant-level impression using transfer copings and polyvinyl siloxane material.
  Arms: Closed-Tray Conventional Impression

SUMMARY:
This prospective controlled clinical trial evaluates the three-dimensional positional accuracy of implant-level impressions obtained using scannable healing abutments compared with conventional open-tray and closed-tray impression techniques in partially edentulous patients with unilateral free-end saddle situations.

DETAILED DESCRIPTION:
Accurate transfer of implant position is critical for achieving passive fit of implant-supported prostheses. This study compares the trueness of implant impressions obtained using a digital workflow based on scannable healing abutments with conventional open-tray and closed-tray impression techniques. Twenty-two partially edentulous patients with unilateral distal extension ridges will undergo all three impression techniques. Three-dimensional deviations will be quantified using best-fit superimposition and root mean square analysis, with the open-tray technique serving as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patients with unilateral free-end saddle (Kennedy Class II)
* Adequate bone for two implants
* Good systemic health
* Ability to provide informed consent

Exclusion Criteria:

* Active periodontal disease
* Poor oral hygiene
* Parafunctional habits
* Temporomandibular disorders
* Heavy smoking (>10 cigarettes/day)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Three-dimensional implant positional accuracy (RMS deviation) | Periprocedural (single assessment, 1 week after second-stage implant surgery)
  Root mean square (RMS) deviation (µm) between test impressions and the open-tray reference model using 3D metrology software.

SECONDARY OUTCOMES:
Comparison of implant positional accuracy between impression techniques | Periprocedural (single assessment, 1 week after second-stage implant surgery)
  Pairwise comparison of RMS deviation values among scannable healing abutment, open-tray, and closed-tray impression techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. The data generated in this study include identifiable clinical and radiographic measurements that are specific to the study protocol and participants. De-identified aggregate data are reported in the published manuscript.